CLINICAL TRIAL: NCT06264609
Title: Novel Precision Medicine Approach to Treatment of Osteoporosis Based on Bone Turnover - Follow Up Study
Brief Title: Precision Medicine Approach for Osteoporosis - Follow Up Study
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Paul F Netzel (Other)
Responsible Party: Sponsor-Investigator, Paul F Netzel, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 91026
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate; Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 Low Turnover - crossover (Experimental): Alendronate
  Interventions: Drug: Alendronate
- Group 2 Low Turnover - crossover (Experimental): Teriparatide
  Interventions: Drug: Teriparatide
- Group 2 Low Turnover - continuation (Experimental): Alendronate
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Alendronate — Participants in Group 1 low turnover, who have received Teriparatide in the main trial and if it is determined that the participant did not respond well to therapy; will be assigned to Alendronate for 12 months.
  Other Names: Grp 1
  Arms: Group 1 Low Turnover - crossover
Drug: Teriparatide — Participants in Group 2 low turnover who received Alendronate in the main trial and if it is determined that the participant did not respond well to therapy; will be assigned to Teriparatide for 12 months.
  Other Names: Grp 2
  Arms: Group 2 Low Turnover - crossover
Drug: Alendronate — Participants in Group 2 low turnover who received Alendronate in the main trial and if it is determined that the participant responded to therapy; will be continue on Alendronate for 12 months.
  Other Names: Grp 2c
  Arms: Group 2 Low Turnover - continuation

SUMMARY:
Osteoporosis is a health problem of major proportions. It affects more than 40 million Americans and results in more than 2 million fractures annually among Medicare patients alone. Hospital admissions for osteoporotic fractures exceed those of heart attacks, strokes and breast cancer combined. Osteoporosis is commonly considered a disease associated with menopause. This estrogen deficiency related bone loss is characterized by high bone turnover with increased resorption without commensurate changes in bone formation. It is in contrast to age-related bone loss, which starts as early as in the fourth decade of life and continues with increasing age. Age-related bone loss is usually associated with lower bone turnover and decreased bone formation is the main abnormality.

Current therapies do not address age-related bone loss and the special needs of the age-related osteoporosis population is currently ignored. This is to a great degree due to difficulties associated with the bone biopsy necessary for unequivocal determination of bone turnover status. Thus, the current standard of care relies on starting with an antiresorber, which is of limited effectiveness in age-related osteoporosis, and in fact impedes the effectiveness of the appropriate anabolic medication. In a current ongoing study - Novel precision medicine approach to treatment of osteoporosis based on bone turnover. EIRB#70781; efforts are focused on addressing this particular problem.

Our follow-up study seeks to achieve one specific aim: to compare effectiveness of Alendronate vs Teriparatide after participants have been switched at the end of treatment at year one, to the other drug at year two for the same duration of treatment.

DETAILED DESCRIPTION:
This will be a prospective, longitudinal crossover trial for participants who have completed therapy in the main trial - Novel precision medicine approach to treatment of osteoporosis based on bone turnover. EIRB#70781.

Participants will be informed of the continuation / follow-up study at enrollment into the main trial. Participants will be approached for further participation in the continuation trial near the end of the initial 12 months treatment period. Consent will be obtained at the final visit of the main trial and crossover therapy will be initiated at that time.

Participants in Group 1 low turnover, who have received Teriparatide in the main trial and if it is determined that the participant did not respond well to therapy; will be assigned to Alendronate for 12 months. Participants in Group 2 low turnover who received Alendronate in the main trial and if it is determined that the participant did not respond well to therapy; will be assigned to Teriparatide for 12 months. Participants in Group 2 low turnover who received Alendronate in the main trial and if it is determined that the participant responded to therapy; will be continued on Alendronate for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed Osteoporosis by DXA (BMD t-score = -2.5 with or without fragility fractures)
2. Prior enrollment and completion of therapy in the "Novel precision medicine approach to treatment of osteoporosis based on bone turnover" trial.3) Premenopausal, menopausal, and post-menopausal females.
3. 45 years old and older.
4. Normal levels of Vitamin D
5. Absence of all exclusion criteria on clinical workup. Patients diagnosed as osteoporotic due to the presence of

Exclusion Criteria:

1. Pregnant or trying to become pregnant or are breastfeeding
2. Use of systemic anticoagulation (blood thinner)
3. Planned or anticipated oral surgery within the next 12 months
4. Planning to move out of the area within 18 months of the study
5. Inability to stand or sit upright for at least 30 minutes
6. Chronic alcoholism and/or drug addiction
7. Prior radiation therapy (external beam or implant radiation) involving the skeleton (only if randomized to the bone forming drug (anabolic Forteo®))
8. Systemic illnesses or organ diseases that may affect bone (except type 1 or type 2 diabetes mellitus)
9. Clinical condition that may limit study participation (e.g., heart diseases (unstable angina), lung diseases (severe COPD), other infections)
10. Abnormalities of the esophagus (tube connecting the mouth to the stomach) which delay esophageal emptying such as stricture (narrowing) or achalasia (a condition that prevents normal swallowing)
11. Have other bone diseases that are not linked to age or menopause
12. Have a history of malignancy (cancer), not including non-melanoma skin cancer.
13. Vitamin D (Calcidiol) level below the normal range (below 20ng/mL).

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in bone loss | 12 months
  The primary endpoint for the follow up study will be bone loss as determined by the percent change in DXA absolute values of the lumbar spine, femoral neck, total hip and radius measured at baseline, at the end of the one-year trial; and at end of the one year follow up study. DXA is chosen because of its wide availability, low radioactivity exposure, and clinical use.

SECONDARY OUTCOMES:
Percent change in Bone Mass Density at the hip | 12 months
  Secondary endpoints will be percent change in BMD at the hip measured at baseline, at the end of the one-year trial; and at end of the one year follow up study. DXA is chosen because of its wide availability, low radioactivity exposure, and clinical use.

OTHER OUTCOMES:
Trabecular bone score (TBS) | 12 months
  A measure of trabecular texture derived from lumbar spine DXA images measure of trabecular texture derived from lumbar spine DXA images which predicts fracture independently of BMD. TBS is calculated as the slope of the log-log transform of the 2D variogram, where the slope characterizes the rate of gray-level amplitude variations. A steep variogram slope with a high TBS value is associated with better bone structure, whereas low TBS values indicate worse bone structure.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Netzel, DNP, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No